CLINICAL TRIAL: NCT02888522
Title: Pre-emptive Immunomodulation After Allogeneic Stem Cell Transplantation in AML
Acronym: IMODLAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 15-182
Record Dates: First submitted 2016-08-26; First posted 2016-09-05 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2016-08

CONDITIONS: AML
MeSH Terms: interventions — Immunomodulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: immunomodulation — Immunomodulation depending on chimerism

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is now an effective treatment of Acute Myeloid Leukemia (AML). After allo-HSCT, relapses are the major cause of mortality and occur in about 30% of cases. The occurrence of relapses is important during the first three months post-allogeneic transplant, then gradually decreases during the first year post-allograft and then becomes weaker. After relapse, therapeutic options include the reduction of immunosuppression, the administration of donor lymphocytes (DLI), chemotherapy or a new transplant. The performance is influenced by the early introduction of treatment whose effectiveness is related to the importance of tumor burden. Immunomodulation of preemptive strategies have recently been established by decreasing immunosuppression and achieve DLIs in patients with a high risk of relapse, before the occurrence of relapse.

The aim of this study is to evaluate the incidence of relapse following the recommendations of post-allogeneic transplant immunomodulation of the French society of bone marrow transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia
* Allogeneic stem cell transplantation (related or unrelated)

Exclusion Criteria:

* Age under 18 years
* Cord blood transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of recipient chimerism | 3 months
  whole blood chimerism

SECONDARY OUTCOMES:
Percentage of relapse at 1 year | Relapse rate at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, France